CLINICAL TRIAL: NCT04693871
Title: Effect of Left Atrial Appendage Velocity on Left Atrial Structure and Function After Radiofrequency Ablation Combined With Left Atrial Appendage Occlusion.
Status: Completed | Type: Observational
Sponsor: The Second Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Ruiqin xie, Director of the Department of Cardiology in the Second Hospital of Hebei Medical University, The Second Hospital of Hebei Medical University
Other Study IDs: XieRuiqinLAAEV
Record Dates: First submitted 2020-12-10; First posted 2021-01-05 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2020-01

CONDITIONS: Left Atrial Appendage Velocity; Left Atrial Structure; Left Atrial Function
MeSH Terms: interventions — Left Atrial Appendage Closure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- high-flow rate group
  Interventions: Device: Transesophageal ultrasound
- low-flow rate group
  Interventions: Device: Transesophageal ultrasound

INTERVENTIONS:
Device: Transesophageal ultrasound — Patients with nonvalvular atrial fibrillation underwent radiofrequency ablation combined with left atrial appendage closure and recovered to sinus rhythm after the operation. To study the changes of left atrial organization and function of two groups of patients with different left atrial appendage emptying speeds.
  Other Names: Radiofrequency ablation of atrial fibrillation combined with left atrial appendage closure

SUMMARY:
Radiofrequency ablation of atrial fibrillation combined with left atrial appendage closure can not only improve symptoms in patients with non-valvular atrial fibrillation, but also prevent left atrial appendage thrombosis. The safety and effectiveness of left atrial appendage occlusion have been confirmed by randomized controlled trials and actual experience. Among patients with different left atrial appendage emptying speeds, there are limited studies on the structure and function of the left atrial appendage after LAA closure. In this study, patients with persistent nonvalvular atrial fibrillation were selected for radiofrequency ablation combined with LAA closure. The sinus rhythm was restored after the operation. According to the different emptying speed of the left atrial appendage, they were divided into a high-flow rate group and a low-flow rate group. The differences in the structure and function of the left atrium between the two groups were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received atrial fibrillation radiofrequency ablation combined with left atrial appendage closure.

Exclude Criteria

* Patients with incomplete data.
* Device embolism.
* Residual shunt around the device found by transesophageal echocardiography greater than 5 mm.
* Mitral valve stenosis.
* Artificial valve.
* Atrial septal defect.
* Dilated cardiomyopathy
* Moderate Severe mitral regurgitation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-valvular atrial fibrillation between the ages of 18 and 80 received atrial fibrillation radiofrequency ablation combined with left atrial appendage occlusion, and recovered to sinus rhythm after the operation. According to the different left atrial appendage emptying speed, it is divided into a higher left atrial appendage emptying speed group and a lower left atrial appendage emptying speed group.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Changes in the structure of the left atrium | 1year
  Measure the left atrial transverse diameter, anteroposterior diameter, upper and lower diameter.
Changes in the function of the left atrium | 1year
  Left atrium volume. Two-chamber and four-chamber left atrium strain and strain rate, left atrium storage function, channel function and pump function.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No